CLINICAL TRIAL: NCT00004203
Title: A Phase II Study of Oxaliplatin in Urothelial Cancer
Brief Title: Oxaliplatin in Treating Patients With Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10020; UCCRC-10020; NCI-T99-0009
Record Dates: First submitted 2000-01-21; First posted 2004-02-12 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): On Day 1 of each 21-day treatment cycle, patients receive 130 mg/m2 oxaliplatin diluted in 250 to 500 mL Dextrose 5% in Water infused intravenously over 2 hours through a peripheral or central vein
  Interventions: Drug: oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating patients who have metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, duration of response, and overall survival of patients with metastatic urothelial carcinoma treated with oxaliplatin. II. Determine the toxicity, including objective measurement of neurotoxicity, of oxaliplatin in these patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified by platinum therapy status (platinum sensitive vs platinum resistant). Patients receive oxaliplatin IV over 2 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression, other illness that would preclude administration of study drug, or unacceptable toxicity. Patients are followed for a minimum of 2 years or until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven metastatic urothelial carcinoma Bidimensionally measurable disease Platinum sensitive OR platinum resistant Platinum sensitive disease: No prior platinum containing regimen OR Progressive or recurrent disease more than 6 months after responding to a platinum containing regimen Platinum resistant disease: Progressive or recurrent disease within 6 months of a platinum containing regimen (cisplatin or carboplatin) No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT or SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance at least 30 mL/min Cardiovascular: No uncontrolled concurrent illness including, but not limited to: Symptomatic congestive heart failure Unstable angina pectoris Cardiac arrhythmia Other: No clinical evidence of neuropathy worse than grade 1 Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No allergy to platinum compounds or antiemetics No uncontrolled concurrent illness including, but not limited to, an active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent colony stimulating factors during the first course of study therapy Chemotherapy: See Disease Characteristics One prior chemotherapy regimen for metastatic disease allowed Prior neoadjuvant or adjuvant chemotherapy regimen allowed if the interval between this therapy and the first therapy for metastatic disease was at least 6 months At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified Other: No other concurrent investigational agents No HIV positive patients receiving antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-02; Primary Completion 2002-02 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Response Rate of Metastatic Urothelial cancer to a single agent oxaliplatin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (14):
- United States (11):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Evanston Northwestern Health Care, Evanston, Illinois
  - Division of Hematology/Oncology, Park Ridge, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
- Canada (3):
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario